CLINICAL TRIAL: NCT04633460
Title: Acute Effects of Exogenous Ketone Ester Administration in Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Kenneth B Margulies, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 833870
Record Dates: First submitted 2020-10-23; First posted 2020-11-18 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Intervention Model Description: Overview: The overall study design will be a randomized, double-blind crossover comparison of ketone ester (KE) therapy vs. KE-free vehicle in 20 patients with established HF with preserved ejection fraction (HFpEF). The main outcomes will be measures of exercise performance (peak and submaximal exercise).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketone ester (Experimental): (R)-3-hydroxybutyl (R)-3-hydroxybutyrate, a ketone ester
  Interventions: Dietary Supplement: Ketone ester
- Placebo (Placebo Comparator): KE-free solution
  Interventions: Dietary Supplement: placebo drink

INTERVENTIONS:
Dietary Supplement: Ketone ester — A nutraceutical ketone ester (KE), (R)-3-hydroxybutyl (R)-3-hydroxybutyrate which provides systemic ketosis
  Arms: Ketone ester
Dietary Supplement: placebo drink — KE free placebo drink
  Arms: Placebo

SUMMARY:
The purpose of this study is to test whether a ketone ester drink will improve exercise in people with heart failure (HF) compared to a placebo. In HF, patients are limited in their ability to do all the things they want to do, and exercise as much as they would like, due to becoming tired and short of breath early. There may be several reasons why these symptoms occur.

There is some evidence that in addition to problems with the heart, patients with HF also have problems with their arteries and muscles that affect their ability to exercise. Ketones have been shown to improve exercise capacity in healthy volunteers, which may be related to effects on the heart function or on muscles. An infusion of ketones through an intravenous (IV) line has also been shown to significantly improve heart function, but whether a drink can produce similar improvements in HF patients is not known. This drink has been given status by Food and Drug Administration as "generally regarded as safe".

The use of DeltaG in this study is experimental. DeltaG has not been approved by the Food and Drug Administration (FDA) for the use being evaluated in this study.

DETAILED DESCRIPTION:
This is a randomized, crossover trial of ketone ester versus placebo in 20 patients with heart failure with preserved ejection fraction. Participants come for a baseline assessment. If they meet eligibility criteria, they are randomized to receive ketone ester first or placebo first. After approximately a week washout period, participants return for the last visit to receive the product they did not receive at the previous visit.

ELIGIBILITY:
Inclusion criteria:

1. Left ventricular ejection fraction ≥ 50%
2. Evidence for elevated filling pressures as follows (at least one of the following between a-d):

   a. Mitral early (E)/mitral septal tissue annular (e') velocity ratio > 8 in addition to one of the following: i. Large left atrium (LA>4.0 cm width or LA volume index >34 mL/m2) ii. Chronic loop diuretic use for control of symptoms iii. Elevated natriuretic peptides within the past year (NT-proBNP>125 pg/ml or BNP>35 pg/ml) b. Mitral E/e' ratio > 14 at rest or with exercise c. Elevated invasively-determined filling pressures previously (resting left ventricular end-diastolic pressure >16 mm Hg or pulmonary capillary wedge pressure > 15 mmHg; or PCWP/LVEDP ≥ 25 mmHg with exercise) d. Prior episode of acute heart failure requiring IV diuretics with evidence of volume overload on exam/radiology or elevated natriuretic peptides.

Exclusion Criteria

1. Intentional ketogenic (high fat, low carbohydrate) diet in the last week or use of ketogenic medications (SGLT2 inhibitors)
2. Significant liver disease (liver function tests > 3x upper limit of normal, cirrhosis) or alcohol abuse disorder (>14 drinks/week).
3. Contraindications to stress testing, conditions that limit exercise, and other clinically-significant causes of exertional limitation (claudication with peripheral artery disease, atrial fibrillation and heart rate >110 at rest, systolic blood pressure>180 mmHg or diastolic blood pressure>110 mmHg, infiltrative/hypertrophic/inflammatory cardiomyopathy, clinically significant pericardial disease, joint or neuromuscular disease that precludes exercise, acute coronary syndrome within the last 2 months, estimated glomerular filtration rate<30 mL/min/1.73 m2, and hemoglobin < 9 mg/dL).
4. Clinically significant lung disease. This would be defined by severe obstructive lung disease (Gold stage 3), a requirement for supplemental oxygen, or chronic obstructive pulmonary disease with an exacerbation requiring steroids or antibiotics within the last 2 months.
5. >= Moderate aortic stenosis, >mild mitral stenosis, >= moderate aortic or mitral regurgitation on screening echocardiogram
6. Type 1 diabetes mellitus
7. Pregnant women. Due to unknown affects of nutritional ketosis in pregnant women, pregnancy will be an exclusion. Accordingly, women of childbearing age with a menstrual cycle within the past year will be asked to submit a urine specimen for pregnancy testing.
8. Angina due to epicardial coronary disease or known presence of clinically-significant, unrevascularized epicardial coronary disease, in the investigator's opinion.
9. Prior reduced LVEF to < 45%

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Selvaraj S, Karaj A, Chirinos JA, Denney N, Grosso G, Fernando M, Chambers K, Demastus C, Reddy R, Langham M, Kumar D, Maynard H, Pourmussa B, Prenner SB, Cohen JB, Ischiropoulos H, Rickels MR, Poole DC, Church DD, Wolfe RR, Kelly DP, Putt M, Margulies KB, Zamani P. Crossover Trial of Exogenous Ketones on Cardiometabolic Endpoints in Heart Failure With Preserved Ejection Fraction. JACC Heart Fail. 2025 Dec;13(12):102435. doi: 10.1016/j.jchf.2025.03.002. Epub 2025 Mar 29. PMID 40243975

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 26 consented participants, 5 screen failed and 1 participant withdrew, leading to 20 randomized participants.
Groups:
- Ketone Ester First, Then Placebo: (R)-3-hydroxybutyl (R)-3-hydroxybutyrate, a ketone ester
  Ketone ester: A nutraceutical ketone ester (KE), (R)-3-hydroxybutyl (R)-3-hydroxybutyrate which provides systemic ketosis.
  10 individuals were randomized to acute dosing of KE first. Then, after approximately 7 day washout, these 10 individuals received acute dosing of placebo.
- Placebo First, Then Ketone Ester: KE-free solution first, then KE after 7 day washout
  placebo drink: KE free placebo drink
  10 individuals were randomized to acute dosing of placebo first. Then, after approximately 7 day washout, these 10 individuals received acute dosing of KE.
Period: First Intervention
Arm/Group | Ketone Ester First, Then Placebo | Placebo First, Then Ketone Ester
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout
Arm/Group | Ketone Ester First, Then Placebo | Placebo First, Then Ketone Ester
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Ketone Ester First, Then Placebo | Placebo First, Then Ketone Ester
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 20 randomized participants are included.
Groups:
- Randomized First to Ketone Ester: (R)-3-hydroxybutyl (R)-3-hydroxybutyrate, a ketone ester
  Ketone ester: A nutraceutical ketone ester (KE), (R)-3-hydroxybutyl (R)-3-hydroxybutyrate which provides systemic ketosis.
  10 individuals were randomized to ketone ester first, and 10 individuals were randomized to placebo first.
- Randomized First to Placebo: KE-free solution
  placebo drink: KE free placebo drink.
  10 individuals were randomized to ketone ester first, and 10 individuals were randomized to placebo first.
- Total: Total of all reporting groups
Arm/Group | Randomized First to Ketone Ester | Randomized First to Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (7) | 71 (10) | 71 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximal Exercise Capacity (Peak VO2) Assessed by Cardiopulmonary Exercise Testing
Description: Peak VO2
Time Frame: Assessed 60 minutes after the intervention.
Population: All 20 participants contributed to the data. 10 participants started first in the ketone ester group and then crossed over to placebo, while 10 participants started first in the placebo arm and crossed over the ketone ester.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Ketone Ester | Placebo
Number analyzed (Participants) | 20 | 20
L/min | 1.0 (0.3) | 1.0 (0.3)

2. Primary Outcome: Submaximal Exercise Capacity (Exercise Time at 75% of Peak Workload) Assessed by Cardiopulmonary Exercise Testing.
Description: Exercise time at 75% of peak workload
Time Frame: Assessed 30 minutes after the intervention.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ketone Ester | Placebo
Number analyzed (Participants) | 20 | 20
minutes | 9.7 (7.3) | 8.7 (4.3)

3. Secondary Outcome: Percent Change in Systemic Vascular Resistance With Exercise
Description: Percent change in systemic vascular resistance with exercise
Time Frame: Assessed 60 minutes after the intervention.
Population: All participants with available data (13 in ketone ester group and 14 in the placebo group) shown here.
Measure: Mean (Standard Deviation); unit: Percent change from rest to peak exercis
Arm/Group | Ketone Ester | Placebo
Number analyzed (Participants) | 13 | 14
Percent change from rest to peak exercis | -21.5 (14.7) | -34.2 (11.5)

4. Secondary Outcome: Substrate Utilization (Reflected by the Respiratory Exchange Ratio) Assessed by Cardiopulmonary Exercise Testing.
Time Frame: Assessed 60 minutes after the intervention.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Ketone Ester | Placebo
Number analyzed (Participants) | 20 | 20
Ratio | 1.09 (0.13) | 1.14 (0.14)

5. Secondary Outcome: VO2 Efficiency (Total Work Performed Over Oxygen Consumed) During Submaximal Cardiopulmonary Exercise Testing.
Time Frame: Assessed 60 minutes after the intervention.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kJ/L O2
Arm/Group | Ketone Ester | Placebo
Number analyzed (Participants) | 20 | 20
kJ/L O2 | 6.0 (2.6) | 6.1 (2.9)

6. Secondary Outcome: Presence of Exercise-induced Arrhythmias (Significant Atrial or Ventricular Arrhythmias)
Time Frame: Assessed throughout the study visit date after the intervention is given (until leaving the research study center that day).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ketone Ester | Placebo
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected the day of the study visit (the day of the first intervention visit, "Day 1", and the day of the second intervention visit, approximately "Day 8").
Arm/Group | Ketone Ester | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 7/20 | 6/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketone Ester (N=20) | Placebo (N=20)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketone Ester (N=20) | Placebo (N=20)
Dizziness (Nervous system disorders) | 3 | 1
Reflux (Gastrointestinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Knee pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Hematoma (Blood and lymphatic system disorders) | 1 | 1
Hypotension (Cardiac disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1
Heart racing (Cardiac disorders) | 0 | 1
Pain with blood draw (Blood and lymphatic system disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT04633460/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT04633460/SAP_001.pdf